CLINICAL TRIAL: NCT00383825
Title: Interventional Study of Vascularization Detected by ICG Angiography in Amniotic Membrane Graft and Conjunctival Autograft After Pterygium Excision
Brief Title: ICG Angiography in Amniotic Membrane Graft and Conjunctival Autograft After Pterygium Excision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: B02-123456-2
Record Dates: First submitted 2006-10-02; First posted 2006-10-04 (Estimated); Last update posted 2006-10-04 (Estimated); Status verified 2006-10

CONDITIONS: Pterygium
Keywords: conjunctival autografts; amniotic membrane; indocyanine green angiography; pterygium surgery
MeSH Terms: conditions — Pterygium

INTERVENTIONS:
Procedure: Anterior segment indocyanine green angiography

SUMMARY:
To evaluate graft vascularization and compare the vascularization patterns of conjunctival autografts with amniotic membrane grafts to better understand the factors involved in pterygium recurrence.

DETAILED DESCRIPTION:
The vascularization and perfusion of conjunctival autografts and amniotic membrane grafts after surgery may have significance in terms of pterygium recurrence and progression. Fluorescein angiography of the anterior ocular segment has been used to evaluate ocular inflammation in scleral inflammation. However, when fluorescein is used, the quality of the angiograms is limited by rapid extravasation of the dye due to diffusion through the fenestrated capillaries of the conjunctiva and episclera. Because fluorescein has a low molecular weight and is not a protein bound molecule, patchy leakage during the first transit of the dye, which obscures the angiographic details even before the late phases of the angiogram, can be seen.

In contrast, indocyanine green (ICG) is a larger molecule than fluorescein and is more highly found in protein bound form. Therefore, it remains within the fenestrated vessels and shows negligible extravasation, which makes it ideal for use in anterior segment angiography.

Tan and coworkers have shown that the morphology of pterygium recurrence inevitably reflects a high degree of vascularity.

In this prospective study, we evaluated the anterior segment indocyanine green angiography (ICGA) findings for graft vascularization after primary pterygium excision with LCAT or AMT.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had primary pterygium

Exclusion Criteria:

* Patients with major systemic diseases (eg, diabetes), vascular disease (excluding hypertension), serious ocular surface disease (eg, cicatricial pemphigoid), glaucoma and previous history of ocular surgery
* Patients with pterygia of both eyes

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 2003-01; Study Completion 2004-12

PRIMARY OUTCOMES:
After intravenous injection of ICG dye, photographs were taken at approximately 1- to 2-second intervals until the first appearance of the dye, and then at 10-second intervals for the next 4 minutes.
Thereafter, photographs were captured at 5, 10, and 20 minutes.
ICGA results of all patients were evaluated at monthly intervals after surgery.
Showing the re-vascularization during the follow-up period was the primary measure.

CONTACTS AND LOCATIONS:
Overall Officials: Yonca A Akova, Md, Study Director — Bakent University Faculty of Medicine Department of Ophthalmology
Locations (1):
- Baskent University Hospital Department of Ophthalmology, Ankara, Turkey (Türkiye)